CLINICAL TRIAL: NCT06239506
Title: Exposure to Novel Brominated and Organophosphate Flame Retardants and Associations With Type 2 Diabetes
Brief Title: Novel Brominated and Organophosphate Flame Retardants and Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiaoling Guan (Other)
Responsible Party: Sponsor-Investigator, Xiaoling Guan, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2021-064-1
Record Dates: First submitted 2023-12-11; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes; Novel Brominated Flame Retardants; Organophosphate Flame Retardants; Fasting Plasma Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples were collected in vacutainer tubes without anticoagulants. The levels of FPG, TG, TC, HDL-C, and LDL-C were measured at the above hospital. The whole blood samples in tubes were centrifuged at 4 000 r min-1 for 10 min, and were placed in two sample tubes. One n was used for determination of FPG and lipid fractions in the hospital. And the other was maintained at -20 ℃ for FRs analysis. FPG was determined enzymatically, and lipid fractions were analyzed using an enzymatic spectrophotometric method in serum . Total lipids (TLs) were counted using Phillip's formula: TL = 2.27 × TC + TG + 0.623.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- type 2 diabetes: Case group participants were recruited from patients diagnosed with type 2 diabetes and undergoing medical treatment at the First Affiliated Hospital of Shandong First Medical University(Shandong Provincial hospital)
  Interventions: Other: no intervention
- Control group: Control group participants were recruited from residents living in Jinan and undergoing physical examinations at the same hospital.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
As alternative flame retardants (FRs), novel brominated flame retardants (NBFRs) and organophosphate flame retardants (OPFRs) are ubiquitous in environment and may cause endocrine disruption effects. The associations between traditional endocrine-disrupting chemicals (EDCs) and type 2 diabetes have been extensively reported in epidemiological studies. To date, however, human-based evidence on the effects of NBFRs and OPFRs is lacking. The investigators conducted a case-control study of 344 participants aged 25-80 years from Shandong Province, East China, to assess potential associations between serum NBFR and OPFR concentrations and etiology of type 2 diabetes for the first time.

DETAILED DESCRIPTION:
In this study, the investigators conducted a case-control study in Shandong Province, East China, to evaluate the associations between serum NBFR and OPFR and risk of type 2 diabetes. The aims of the present study were to (1) evaluate the associations between alternative FRs in human serum and the risk of type 2 diabetes, (2) assess the relationships between alternative FR concentrations and fasting plasma glucose (FPG), (3) investigate the correlations between alternative FRs and concentrations of lipid fractions, including TG, TC, high-density lipoprotein cholesterol (HDL-C), and low-density lipoprotein cholesterol (LDL-C), and (4) clarify the joint effects of NBFR and OPFR mixtures on the risk of type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

Group of Type 2 diabetes patients:

1. age 18 ~ 75 years old;
2. type 2 diabetes patients diagnosed in the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province) , HBA1C ≥7.0% and <10.5% ;
3. patients signed informed consent.

Control Group:

1. age 18 ~ 75 years old;
2. healthy population recruited from the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province) ;
3. living in the monitoring area for more than 6 months within 12 months;
4. normal thyroid function and no history of thyroid cancer were needed in the control group;
5. Fasting Blood Glucose level of 0.7 mmol/l was needed in the Control Group of Type 2 diabetes Mellitus Without History of diabetes;
6. patients with informed consent.

Exclusion Criteria:

* Group of Type 2 diabetes:

  1. pregnant, lactating women, patients with acute cardiac cerebrovascular disease;
  2. patients with severe liver and Renal Impairment (related laboratory tests more than 2 times the normal) ;
  3. patients with Type 1 diabetes;
  4. participants in other clinical trials within 3 months;
  5. patients with malignant tumors.
  6. has the disease and so on serious anemia, is not suitable to carry on the patient which the blood draws the test.

Control Group:

1. patients with serious heart, liver or kidney disease;
2. patients with iodine or Thyroid hormone;
3. patients with confirmed malignant tumor;
4. pregnant women or those who have recently taken contraception or estrogen.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: we will conduct a case-control study of 340 participants from Shandong 116 Province, East China, to evaluate the associations between serum NBFR and OPFR and risk of type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
alternative FRs | 2022.1-2024.12
  Determination of FRs was performed by a gas chromatography triple quadrupole mass spectrometry (GC-MS/MS, TQ-8050NX, Shimadzu, Japan) equipped with an electron ionization (EI+) ion source.

SECONDARY OUTCOMES:
levels of FPG | 2022.1-2024.12
  Detecting blood sugar using a biochemical analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Tian Hui, Dr., Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided